CLINICAL TRIAL: NCT00771004
Title: Pilot Trial Studying the Effects of Pioglitazone in Comparison to Placebo on Myocardial Function and Oxidative Stress in Patients With Type II Diabetes and Insulin Resistance Undergoing Elective PTCA. A Randomized Double-blinded Phase II Study.
Brief Title: Efficacy of Pioglitazone on Myocardial Function in Patients Undergoing Coronary Stent Implantation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Pharma GmbH, Aachen (Germany)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATS K021; 2006-002237-20 (EudraCT Number); D-PIO-111 (Other: Takeda ID); U1111-1115-9160 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Oxidative Stress; Coronary Artery Disease; Type 2 Diabetes
Keywords: drug effects; Type II Diabetes; Angioplasty, Transluminal, Percutaneous Coronary; Drug Therapy; Heart; physiology; function
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone 30 mg to 45 mg QD (Experimental)
  Interventions: Drug: Pioglitazone
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 30 mg, tablets, orally, once daily for one week; increased to Pioglitazone 45 mg, tablets, orally, once daily for up to two weeks.
  Other Names: ACTOS®; AD4833
  Arms: Pioglitazone 30 mg to 45 mg QD
Drug: Placebo — Pioglitazone placebo-matching tablets, orally, once daily for up to three weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the effects of pioglitazone, once daily (QD), on heart functioning before, during and after stent implantation.

DETAILED DESCRIPTION:
Type 2 diabetes increases the risk of coronary heart disease at least by two to three fold compared with non-diabetic subjects. Moreover, prospective studies have shown a significant correlation between several glycemic confounders and morbidity from coronary heart disease even in patients without diabetes mellitus. In patients with previously diagnosed coronary heart disease, impaired glucose tolerance was found in 30 to 67 %. The cardiovascular risk of patients with insulin resistance, with or without glucose intolerance has become more and more apparent within recent years and quantitative coronary angiographic studies have revealed a correlation between the severity of coronary heart disease and impaired glucose tolerance.

A new pharmaceutical class for the intervention of insulin resistance, the peroxisome proliferator activated receptor (gamma) agonists have been successfully introduced in the treatment of type 2 diabetes. Beyond their metabolic effects on glucose and lipid metabolism, peroxisome proliferator activated receptor (gamma) agonists show to exert a couple of pleiotropic, anti-inflammatory and vasoprotective effects in patients with type 2 diabetes and impaired glucose tolerance.

The incidence and severity of peri-procedural myocardial injury during percutaneous coronary interventions with stent implantation in diabetic and in non-diabetic patients is an important prognostic confounder for the patient. Different laboratory biomarkers have been investigated as diagnostic tools for the estimation of the risk of peri-procedural myocardial injury. Recent studies have convincingly demonstrated that the risk of subsequent ischemic heart events is related to the extent of cardiac troponin or CK-MB increase after coronary intervention, and the prognosis for these individuals is usually worse than that for patients who do not develop an increase in these biomarkers.

In a recent trial it was shown that pretreatment with atorvastatin could reduce procedural myocardial injury in elective coronary intervention. The incidence of Troponin I increase was 48% in the placebo group compared to 20% in the atorvastatin group.

The aim of this study is to investigate the effect of pioglitazone on the incidence of peri-procedural myocardial injury in patients undergoing percutaneous coronary interventions with stent implantation. Total participation time is anticipated to be 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary artery disease with planned percutaneous coronary intervention with stent implantation.
* Type II-diabetics and/or an IRIS II score greater than or equal to 50 (measure for the identification of patients with insulin resistance and increased vascular risk).
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* A planned percutaneous coronary intervention with stent implantation less than 15 days after the screening visit.
* Planned multi-vessel intervention.
* Use of systemic corticosteroids within the last 3 months prior to screening visit.
* Anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structures.
* History of severe or multiple allergies.
* Treatment with any other investigational drug within 3 months before trial entry or earlier participation in the present study.
* Have had more than one unexplained episode of severe hypoglycemia (defined as requiring assistance of another person due to disabling hypoglycemia) within 6 months prior to screening visit.
* Progressive fatal disease.
* History of drug or alcohol abuse within the last 10 years.
* A history of significant cardiovascular (New York Health Association stage II - IV), respiratory, gastrointestinal, hepatic (alanine aminotransferase greater than 2.5 times the normal reference range), renal (creatinine greater than 1.2 mg/dL in women and greater than 1.5 in men and/or glomerular filtration rate less than 45), neurological, psychiatric and/or hematological disease as judged by the Investigator.
* Pre-treatment with peroxisome proliferator-activated receptor (gamma) agonists within the 3 months prior to screening.
* If insulin therapy applicable: initiation of insulin therapy within the last 3 months.
* If statin therapy applicable: change of medication within the last 4 weeks.
* Myocardial infarction within 3 months prior to screening visit.
* Blood donation within last 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Cardiac Troponin I elevation (greater than 1 upper limit of normal) post-percutaneous coronary intervention with stent implantation. | 24 hours post stent implantation.

SECONDARY OUTCOMES:
Incidence of Creatine Kinase (Myocard-type) post-percutaneous coronary intervention with stent implantation. | 24 hours post stent implantation.
Mean peak values of Troponin I and Creatine Kinase (Myocard-type) post-percutaneous coronary intervention with stent implantation. | Hours: 2, 6 and 12 and 24 post stent implantation.
Frequency of Doppler-detected microembolism measured by high intensity transient signals during percutaneous coronary intervention with stent implantation (sub-study Jena only). | Duration of stent implantation surgery.
Time course of Troponin I Laboratory Procedure. | Visits: 2, 3, 4, 5, 6, 7, and 8 or Final Visit.
Time course of high-sensitive-C-Reactive Peptide Laboratory Procedure. | Visits: 2, 3, 4, 5, 6, 7, and 8 or Final Visit.
Time course of nitrotyrosine Laboratory Procedure. | Visits: 2, 3, 4, 5, 6, 7, and 8 or Final Visit.
Time course of Asymmetric dimethylarginine Laboratory Procedure. | Visits: 2, 3, 4, 5, 6, 7, and 8 or Final Visit.
Time course of E-selectin Laboratory Procedure. | Visits: 2, 3, 4, 5, 6, 7, and 8 or Final Visit.
Time course of Myoglobin Laboratory Procedure. | Visits: 2, 3, 4, 5, 6, 7, and 8 or Final Visit.
Time course of Visfatin Laboratory Procedure. | Visits: 2, 3, 4, 5, 6, 7, and 8 or Final Visit.
Time course of Proinsulin intact Laboratory Procedure. | Visits: 1 and 7 or Final Visit.
Time course of Adiponectin Laboratory Procedure. | Visits: 1 and 7 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Adviser Clinical Research, Study Director — Takeda Pharma Gmbh, Aachen (Germany)
Locations (7):
- Germany (7):
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Kassel, Hesse
  - Wiesbaden, Hesse
  - Wuppertal, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Jena, Thuringia

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI